CLINICAL TRIAL: NCT06103019
Title: Comparison of Patient Satisfaction and Chewing Efficiency Between Conventional and 3D Printed Complete Dentures. A Randomized Crossover Clinical Trial
Brief Title: Comparison of Patient Satisfaction and Chewing Efficiency Between Conventional and 3D Printed Complete Dentures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma mahanna (Other)
Responsible Party: Sponsor-Investigator, Fatma mahanna, lecturer of prosthodontics, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A04080120
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: A crossover design was conducted. Each patient received two prostheses: 1) Conventional Maxillary and mandibular complete denture. 2) 3D printed Maxillary and mandibular complete denture.Each denture was used for 3 months followed by 2 weeks rest period without wearing the denture then the other type of denture was delivered and used for another 3 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional (complete denture) (Active Comparator): Each patient received two prostheses: 1) Conventional Maxillary and mandibular complete denture. 2) 3D printed complete Maxillary and mandibular complete denture. The succession of complete denture insertion was randomized to reduce the impact of the order of the complete denture on patient satisfaction outcomes. Each denture was used for 3 months followed by 2 weeks rest period without wearing denture then the other type of denture was delivered and used for another 3 months.
  Interventions: Other: conventional complete denture; Other: 3D complete denture
- 3D printed complete denture (Active Comparator): Each patient received two prostheses: 1) Conventional Maxillary and mandibular complete denture. 2) 3D printed complete Maxillary and mandibular complete denture. The succession of complete denture insertion was randomized to reduce the impact of the order of the complete denture on patient satisfaction outcomes. Each denture was used for 3 months followed by 2 weeks rest period without wearing denture then the other type of denture was delivered and used for another 3 months.
  Interventions: Other: conventional complete denture; Other: 3D complete denture

INTERVENTIONS:
Other: conventional complete denture — conventional complete denture. The succession of complete denture insertion was randomized to reduce the impact of the order of the complete denture on patient satisfaction outcomes. Each denture was used for 3 months followed by 2 weeks rest period without wearing the denture then the other type of denture was delivered and used for another 3 months and vice versa.
Other: 3D complete denture — 3D complete denture. The succession of complete denture insertion was randomized to reduce the impact of the order of the complete denture on patient satisfaction outcomes. Each denture was used for 3 months followed by 2 weeks rest period without wearing the denture then the other type of denture was delivered and used for another 3 months and vice versa.

SUMMARY:
Twenty completely edentulous patients were enrolled in this study. Each patient received two types of prostheses. 1) Conventional complete dentures. 2) 3D printed dimethacrylate-based resin complete dentures. Patient satisfaction was assessed using the oral health impact profile (OHIP-EDENT-N) survey questionnaire, and masticatory performance was evaluated with the two-colored chewing gum mixing ability by evaluation of the standard deviation of hue at (T0) at the time of complete denture insertion, (T3) after 3 months of denture use and (T6) after 6 months of denture use.

DETAILED DESCRIPTION:
For each patient, conventional maxillary and mandibular complete dentures were constructed, followed by 3D printed complete dentures construction as follows: Scanning of maxillary and mandibular complete dentures and scanning of master casts were done using 3D scanner (VDSL Home Gateway model EchoLife DG8045 China) after lightly coated with anti-glare spray (Siladent Marmoscan spray basic Ref. 250022). The resultant data in STL format were transmitted to the CAD-CAM complete denture provider using a purpose-built software program (Exocad DentalIDB 2.4 plovdiv7290[version 2.4 Enginebuld 7290]). The anatomic landmarks were identified, and the peripheral limits were marked on a virtual model in the design software, which then were served to design the definitive complete denture.

The scanned STL image of the conventional complete denture which have been previously constructed was superimposed on the newly designed denture for comparison of polished surface, teeth alignment, size, and form of teeth. A digital preview was generated and sent for approval before fabrication.

Printing Preparation: The denture base shade was selected, and then the cassette of the 3D printer (RASDENT 3D printer) was filled with fresh DENTCA Denture Base II dimethacrylate-based resins with photo-initiator). Then the printer door closed. Printing procedures: The denture base model STL file was uploaded into the software. The denture base was oriented vertically on the build platform. Supports were generated around the perimeter of the denture base. The desired slice thickness was selected and then the printing was started. Cleaning, Bonding teeth to the denture base, Post-curing procedures, Finishing Evaluation of patient satisfaction: The OHRQoL of the patient was assessed using an instrument called OHIP-EDENT-N10.

ELIGIBILITY:
Inclusion Criteria:

* They were healthy, free from any systemic diseases affecting bone metabolism such as uncontrolled diabetics or osteoporosis. This was achieved through detailed medical history and clinical examination by physician. They had no previous denture experience. Residual alveolar ridges covered with healthy firm mucosa. Angle's class I maxilla-mandibular relationship.

Exclusion Criteria:

* Systemic disease

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 months
  The Oral health-related quality of life (OHRQoL) of the patient was assessed using an instrument called OHIP-EDENT-N A simple score was calculated by adding the responses to all the questions (0 = never; 1= seldom; 2 = fairly often; 3 = often; 4 = very often)

SECONDARY OUTCOMES:
chewing efficiency | 6 months
  two-color mixing ability test (colorimetric method)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No